CLINICAL TRIAL: NCT06780475
Title: Validation of in Vitro Method for Anti-MCPyV Immunotherapy on Patients With Merkel Cell Carcinoma of Skin
Brief Title: Validation of in Vitro Method for Anti-MCPyV Immunotherapy on Patients With Cutaneous Merkel Cell Carcinoma
Acronym: VIRASKIN
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP240470; 2024-A00643-44 (Registry Identifier: IDRCB)
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Merkel Cell Carcinoma of Skin
Keywords: Merkel Cell Carcinoma of Skin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to test and validate in vitro a cell therapy approach for MCPyV+ Merkel Cell Carcinoma patients.

DETAILED DESCRIPTION:
The aim of the study is to test and validate in vitro a cell therapy approach for MCPyV+ Merkel Cell Carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years old;
* Diagnosed with Merkel cell carcinoma of skin, ongoing for local treatment, systemic treatment, complementary treatment or an active follow-up;
* Informed for the study and no-opposed for participation;
* Affiliated with a social security scheme or in an equivalent situation.

Exclusion Criteria:

* Patients ongoing another interventional clinical trial;
* Patients under guardianship or trusteeship;
* Pregnancy or breastfeed;
* Patients refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of Merkel cell carcinoma of skin, ongoing for local treatment, systemic treatment, complementary treatment or with an active follow-up beside dermatologist.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Anti-MCPyV functionality | Day 0 and Day 4
  Anti-MCPyV functionality, including cytotoxicity, of T cells obtained after in vitro culture.

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Blom, MD, Principal Investigator — Dermato-oncology Department, Ambroise Paré Hospital, APHP; Yassine Taoufik, MD, PhD, Study Director — U1186 INSERM, PAUL BROUSSE Hospital, APHP
Locations (1):
- Dermato-oncology Department, Ambroise Paré Hospital, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No